CLINICAL TRIAL: NCT02608554
Title: Taichi for Treating Overweight/Obese Adolescent and Young Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Taichi for Overweight/Obese Adolescent and Young Women With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yan Li, Associate seiner physician, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Taichi for PCOS
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary sybdrome; Taichi
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taichi (Experimental): The 24 forms of simplified TCC recommended as the popular health sport by the General Administration of Sport of China were applied.
  Interventions: Behavioral: Taichi
- Self-monitored exercise (Active Comparator): Exercise was self-monitored and consisted of brisk walking, cycling, jogging, or any other aerobic exercise.
  Interventions: Behavioral: Self-monitored exercise

INTERVENTIONS:
Behavioral: Taichi — The program of Taichi training consisted of 60 minutes exercise sessions, 3 days per week for 12 weeks, based on their original level of physical activity. Each session comprised 40 minutes of Taichi training plus a 10-minute warm-up and cool-down. The Taichi training was instructed by the same experienced Taichi instructors who were qualified in the teaching of Taichi. The 24 forms of simplified Taichi recommended as the popular health sport by the General Administration of Sport of China were applied.
  Arms: Taichi
Behavioral: Self-monitored exercise — Exercise was self-monitored and consisted of brisk walking, cycling, jogging, or any other aerobic exercise for 60 mins. 3 days per week for 12 weeks.
  Arms: Self-monitored exercise

SUMMARY:
The present study is a randomized pilot study, overweight/obese adolescent and young PCOS subjects will be assigned into two groups: Taichi arm and control arm. Hormonal profile and metabolic profile will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 19 and 35 years;
* Diagnosis of PCOS according to the modified Rotterdam criteria;
* 2 years after menarche;
* Body mass index (BMI) equal to or greater than 23 kg/m*m.

Exclusion Criteria:

* Administration of other medications known to affect reproductive function or metabolism within the past three months, including oral contraceptives, Gonadotropin-releasing hormone (GnRH) agonists and antagonists, anti androgens, gonadotropins, anti-obesity drugs, Chinese herbal medicines, anti diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, and calcium channel blockers.
* Patients with other endocrine disorder including 21-hydroxylase deficiency, hyperprolactinemia, uncorrected thyroid disease, suspected Cushing's syndrome.
* Patients with known severe organ dysfunction or mental illness.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | 3 months

SECONDARY OUTCOMES:
Fasting plasma glucose (Glu) | 3 months
Fasting insulin (Ins) | 3 months
HOMA-IR | 3 months
  HOMA-IR = fasting insulin concentrations (mIU/L) ×fasting plasma glucose concentrations (mmol/L)/22.5
Testosterone (T) | 3 months
Luteinizing hormone (LH) | 3 months
Follicle stimulating hormone (FSH) | 3 months
Waist/hip ratio | 3 months
Ferriman-Gallwey score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lihui Hou, Bachelor, Study Chair — First Affiliated Hospital of Heilongjiang University Of Chinese
Locations (1):
- First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China

REFERENCES:
- [Derived] Li Y, Peng C, Zhang M, Xie L, Gao J, Wang Y, Gao Y, Hou L. Tai Chi for Overweight/Obese Adolescents and Young Women with Polycystic Ovary Syndrome: A Randomized Controlled Pilot Trial. Evid Based Complement Alternat Med. 2022 Jun 17;2022:4291477. doi: 10.1155/2022/4291477. eCollection 2022. PMID 35754690
- [Derived] Li Y, Peng C, Cao G, Li W, Hou L. Tai chi for overweight/obese adolescent and young women with polycystic ovary syndrome: study protocol for a randomized controlled trial. Trials. 2018 Sep 20;19(1):512. doi: 10.1186/s13063-018-2893-z. PMID 30236149